CLINICAL TRIAL: NCT02868632
Title: A Phase I Study of Immune Checkpoint Inhibition (Anti-CTLA4 and/or Anti-PD-L1) in Combination With Radiation Therapy in Patients With Unresectable and Non-metastatic Pancreatic Cancer
Brief Title: Study of Immune Checkpoint Inhibition With Radiation Therapy in Unresectable, Non-metastatic Pancreatic Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: termination because of low accrual; four subjects enrolled and four screen failures.
Sponsor: NYU Langone Health (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-01317
Record Dates: First submitted 2016-08-08; First posted 2016-08-16 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Pancreatic Cancer
Keywords: Unresectable; Locally Advanced; Non-Metastatic
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — durvalumab; tremelimumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A: MEDI4736 + SBRT (Experimental): MEDI4736 10 mg/kg IV every 2 weeks plus Stereotactic Body Radiation (SBRT) 6 Gy x 5 Days, 10 Subjects
  Interventions: Drug: MEDI4736; Radiation: Stereotactic Body Radiation Therapy (SBRT)
- Cohort B:Tremelimumab + SBRT (Experimental): Tremelimumab 10 mg/kg IV every 4 weeks plus Stereotactic Body Radiation (SBRT) 6 Gy x 5 Days, 10 Subjects
  Interventions: Drug: Tremelimumab; Radiation: Stereotactic Body Radiation Therapy (SBRT)
- Cohort C: MEDI4736 + Tremelimumab + SBRT (Experimental): MEDI4736 + Tremelimumab (recommended phase 2 IV dose for combination) plus Stereotactic Body Radiation (SBRT) 6 Gy x 5 Days, 16 Subjects
  Interventions: Drug: MEDI4736; Drug: Tremelimumab; Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Drug: MEDI4736 — anti-PD-L1 human monoclonal antibody
  Other Names: Durvalumab
  Arms: Cohort A: MEDI4736 + SBRT; Cohort C: MEDI4736 + Tremelimumab + SBRT
Drug: Tremelimumab — anti-CTLA4 human monoclonal antibody
  Other Names: CP-675,206
  Arms: Cohort B:Tremelimumab + SBRT; Cohort C: MEDI4736 + Tremelimumab + SBRT
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Stereotactic body radiation therapy (SBRT) will be administered at the standard dose of 6 Gy daily for 5 days.

SUMMARY:
This is an open-label, three-cohort, phase Ib study to determine the safety, recommended phase 2 dose (RP2D), and efficacy of Stereotactic Body Radiation Therapy (SBRT) in combination with either (A) MEDI4736 alone, (B) tremelimumab alone, or (C) the combination of MEDI4736 and tremelimumab for patients with unresectable locally advanced adenocarcinoma of pancreas.

DETAILED DESCRIPTION:
Patients with unresectable, locally advanced adenocarcinoma of pancreas will receive Stereotactic Body Radiation Therapy (SBRT) at a dose of 6 Gy daily, for 5 days. In Cohort A, where MEDI4736 is given, subjects will receive 10 mg/kg of MEDI4736 every 2 weeks, on the same day as, but after the first dose of SBRT is delivered (within 4 hours). In Cohort B, where tremelimumab is given, subjects will receive 10 mg/kg of tremelimumab every 4 weeks, on the same day as, but after the first dose of SBRT is delivered (within 4 hours). In Cohort C, where MEDI4736 and tremelimumab are given in combination, subjects will receive 10 mg/kg of tremelimumab every 4 weeks, on the same day as, but after the first dose of SBRT is delivered (within 4 hours), followed by 10 mg/kg of MEDI4736 every 4 weeks.

Correlative Studies The investigators will evaluate immune changes in peripheral blood samples and in tumor biopsy fine needle aspirate (FNA) specimens pre- and post- treatment from the 3 cohorts that involve the combination of stereotactic body radiation therapy (SBRT) with either (A) MEDI4736 alone, (B) tremelimumab alone, or (C) the combination of MEDI4736 and tremelimumab. FNA biopsies will be done at baseline (within 30 days of treatment initiation) and Day 28 of cycle 2 (between days 22-28 of cycle 2).

ELIGIBILITY:
Inclusion:

* Histopathological confirmation of pancreatic adenocarcinoma prior to study entry.
* Unresectable and non-metastatic disease
* At least 1 measurable metastatic lesion by RECIST 1.1, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques, or as >10 mm with spiral computed tomography (CT) scan, and that is accessible for biopsy.
* Age >18 years
* ECOG performance status 0-1
* Normal organ and marrow function as defined below:

Absolute Neutrophil Count > 1,000/mcL Platelets ≥ 75,000/mcL Total Bilirubin ≤ 2 x ULN Serum Albumin ≥ 2.5 g/dl ALT or AST up to 3 x ULN if no liver metastases or ALT or AST up to 5 x ULN if liver metastases present Creatinine < 2 x institution upper limit of normal OR Creatinine Clearance > 45 mL/min/1.73 m2, as calculated below, for patients with creatinine levels above institutional normal

* No history of another malignancy in the past 5 years, except for treated non-melanoma skin cancer, superficial bladder cancer, or carcinoma-in-situ of the cervix
* No coexisting medical problems that would limit compliance with the study
* Ability to understand and sign a written informed consent document. Patient must have willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures.
* Female subjects of childbearing potential must have a negative serum pregnancy test prior to study entry
* Female subjects of childbearing potential and males must agree to use a highly effective method of contraception for the duration of study treatment, and for six months after discontinuation of the study drug.

Exclusion:

* Resectable, borderline resectable or metastatic disease
* Prior chemotherapy, targeted therapy, immunotherapy, clinical trials or radiotherapy for pancreatic cancer.
* Active or history of concomitant therapy with any of the following: interleukin (IL) 2, interferon, or other non-study immunotherapy regimens, immunosuppressive agents, other investigational therapies, or chronic use of systemic corticosteroids (inhaled and topical steroids are permitted)
* Active or history of chronic autoimmune disease with symptomatic disease within the 3 years before randomization.
* Active or history of inflammatory bowel disease (colitis, Crohn's disease), irritable bowel disease, celiac disease, or other serious, chronic, gastrointestinal conditions associated with diarrhea.
* Diverticulitis within the past 2 years.
* Active HIV infection
* Uncontrolled systemic disease including, but not limited to, ongoing or active systemic infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Brain metastases
* Patients should not be vaccinated with live attenuated vaccines within 1 month of starting tremelimumab and MEDI4736 treatment.
* History of hypersensitivity reaction to human or mouse antibody products
* Evidence of pre-existing idiopathic pulmonary fibrosis on CT scan at baseline
* Unhealed surgical wound at time of treatment, or history of unhealed surgical wound for more than 30 days
* History of an invasive secondary primary malignancy diagnosed within the previous 3 years, except for appropriately treated stage I endometrial or cervical carcinoma, prostate carcinoma treated surgically or non-melanoma skin cancer.
* Non-protocol antineoplastic agents will not be permitted during this study
* Patients may not recieve other investigational agents.
* Pregnant or lactating women
* Subjects with dementia or significantly altered mental status that would prohibit understanding or rendering of information and consent and compliance with the requirements of the protocol.
* Subjects unable or unwilling to abide by the study protocol or cooperate fully.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08-07 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-03-04 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 24 Months
  Kaplan Meier curves will be used to summarize Overall Survival.

SECONDARY OUTCOMES:
Progression-Free Survival | 24 Months
  Kaplan Meier curves will be used to summarize Progression-Free Survival.
Response Evaluation Criteria in Solid Tumors (RECIST 1.1) | 24 Months
  Response rates will be estimated with exact 95% confidence intervals for each dose level.
Immune-related Response Criteria (irRC) | 24 Hours
  Kaplan Meier curves will be used to summarize Clinical Benefit Rate.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Wu, MD, Principal Investigator — NYU Langone Medical Center
Locations (3):
- United States (3):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - New York University School of Medicine, New York, New York
  - Montefiore Medical Center, The Bronx, New York